CLINICAL TRIAL: NCT07291830
Title: Clinical Effectiveness of a Remineralizing Self-Etch Primer for Orthodontic Bracket Bonding: A Randomized Clinical Trial
Brief Title: A Novel Remineralizing Self-Etch Primer for Orthodontic Bracket Bonding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali I Ibrahim, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1102425
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: White Spot Lesions; Enamel Demineralization
Keywords: Orthodontic Bracket Bonding; Self-Etch Primers

STUDY DESIGN:
Intervention Model Description: Evaluating the clinical effectiveness of enamel etching/priming with M-SEP versus P-SEP in achieving clinically adequate bond strengths throughout the assessment of bracket failure rate over a period of 6 months.
Who Masked: Participant
Masking Description: multi-center, parallel-group, single-blinded randomized clinical trial conducted in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines for orthodontic research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Split-mouth bonding: SEP 1 right/LL vs SEP 2 left/LR (Experimental): Patients receive fixed MBT stainless-steel brackets bonded with two self-etch primers in a split-mouth design. Maxillary right and mandibular left incisors, canines, and premolars are etched with SEP 1; maxillary left and mandibular right counterparts are etched with SEP 2. All teeth are polished with fluoride-free pumice, brackets bonded with Transbond XT, and standard NiTi-stainless-steel archwire sequence used in both arches.
  Interventions: Device: Remineralizing self-etch primer (M-SEP, SEP 1); Device: Standard self-etch primer (P-SEP, SEP 2)
- Split-mouth bonding: SEP 1 left/LR vs SEP 2 right/LL (Experimental): Patients receive the same fixed MBT stainless-steel appliance and archwire sequence as Group A. In this arm, maxillary left and mandibular right incisors, canines, and premolars are etched with SEP 1, while maxillary right and mandibular left counterparts are etched with SEP 2. Bonding follows identical polishing, priming, Transbond XT application, and LED light-curing protocol as in Group A.
  Interventions: Device: Remineralizing self-etch primer (M-SEP, SEP 1); Device: Standard self-etch primer (P-SEP, SEP 2)

INTERVENTIONS:
Device: Remineralizing self-etch primer (M-SEP, SEP 1) — Experimental self-etch primer based on Transbond Plus modified with 7% nano-hydroxyapatite. Applied to labial/buccal enamel of incisors, canines, and premolars after pumice prophylaxis; air-dried 3 s, brackets bonded with Transbond XT and LED light-cured 10 s mesial and 10 s distal.
Device: Standard self-etch primer (P-SEP, SEP 2) — Conventional Transbond Plus self-etch primer used according to manufacturer's instructions for enamel conditioning of incisors, canines, and premolars, followed by Transbond XT adhesive and LED light-curing as above.

SUMMARY:
This randomized clinical trial aims to evaluate the clinical effectiveness of a remineralizing self-etch primer used for orthodontic bracket bonding. The study compares bonding performance, enamel surface effects, and clinical outcomes between the experimental primer and the conventional bonding protocol,verify the potential remineralization effect, and examine the amount of adhesive remnants left on enamel over a period of 6 months.

DETAILED DESCRIPTION:
To evaluate the clinical performance of a newly developed self-etch primer (M-SEP) versus P-SEP in bonding metallic orthodontic brackets to different teeth, verify the potential remineralization effect, and examine the amount of adhesive remnants left on enamel over a period of 6 months.

Objectives:

Primary; Evaluating the clinical effectiveness of enamel etching/priming with M-SEP versus P-SEP in achieving clinically adequate bond strengths throughout the assessment of bracket failure rate over a period of 6 months.

Secondary;

1. Examining the potential enamel remineralization effect of both systems via the use of Fe-SEM and Raman spectroscopy.
2. Assessing the amount of remnant adhesive left post bracket failure (for both systems) via the use of SEM and digital photography.
3. Measuring the total time required for remnant adhesive removal post bracket failure/debonding.
4. Evaluating patient perception during bracket failure/debonding and subsequent adhesive removal procedure.

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition including incisors, canines, premolars, and molars (excepting 3rd molars;
* Teeth with sound, non-carious buccal enamel and no pretreatment with chemical agents such as hydrogen peroxide,
* No previous orthodontic treatment with fixed appliances.

Exclusion Criteria:

* Participants unable to give informed consent,
* Had craniofacial anomalies,
* Require orthognathic surgery as part of their treatment,
* Had congenital enamel defects.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Bracket Bond Failure Rate | 6 MONTH
  Documented as a percentage of brackets debonded during the 6-month observation period, categorized by location (incisor, canine, premolar) and cause (adhesive failure, cohesive failure, bracket fracture .

SECONDARY OUTCOMES:
Adhesive Remnant Index | 6 MONTH
  Adhesive Remnant Index (ARI) scores will be assessed to determine failure mode

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad - Orthodontic Dept/Postgraduate Clinic, Baghdad, Baghdad Governorate, Iraq

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned because patient consent and institutional policy do not allow external sharing of individual-level data."

REFERENCES:
- [Background] Erbe C, Hartmann L, Schmidtmann I, Ohlendorf D, Wehrbein H. A novel method quantifying caries following orthodontic treatment. Sci Rep. 2021 Nov 1;11(1):21347. doi: 10.1038/s41598-021-00561-7. PMID 34725354
- [Background] Garma NMH, Ibrahim AI. Development of a remineralizing calcium phosphate nanoparticle-containing self-etching system for orthodontic bonding. Clin Oral Investig. 2023 Apr;27(4):1483-1497. doi: 10.1007/s00784-022-04767-5. Epub 2022 Nov 2. PMID 36322155